CLINICAL TRIAL: NCT07270926
Title: Feasibility Study of a Patient-centered Clinical Decision Support System for Recommended Screenings in Primary Care
Brief Title: Feasibility Study of a Patient-centered CDS for Recommended Screenings in Primary Care
Acronym: ADER-F
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL23_1126; 2025-A00819-40 (Other: ID-RCB)
Record Dates: First submitted 2025-09-10; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Primary Care
Keywords: Primary care; Recommended screening; Medical Decision Support System (MDSS); patient-centered Clinical Decision Support (CDS)

STUDY DESIGN:
Intervention Model Description: non-comparative experimental feasibility study, in a prospective, multicenter regional phase in the context of primary care clinical practice in France
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADER-F (Experimental): The Lianeli digital platform is a SADM produced by PREVENEAR. The Lianeli SADM is designed to facilitate the identification of patients' eligibility for screening recommended by the HAS (French National Authority for Health), and shared decision-making. It will be used by the patient through a health self-questionnaire and access to factual information sheets, then by the patient and GP during the consultation dedicated to prevention. All the examinations suggested by Lianeli are based on national recommendations, mainly from the HAS.
  A mixed methodology was used, combining the quantitative component with a qualitative component involving semi-structured interviews with volunteer healthcare professionals and a sample of volunteer patients from among those included.
  Interventions: Other: ADER-F quantitative assessment; Other: Individual semi directive interview with the patient; Other: Individual semi directive interview or r Focus Group with the primary care professional

INTERVENTIONS:
Other: ADER-F quantitative assessment — The Lianeli SADM is designed to facilitate the identification of patients eligible for screenings recommended by the HAS (French National Authority for Health) and to facilitate shared decision-making during a primary care consultation dedicated to prevention.
  The Lianeli SADM will be used by the patient first via a health questionnaire, then by the patient and the general practitioner during the consultation dedicated to prevention.
Other: Individual semi directive interview with the patient — 24 Semi-structured individual interviews will be conducted with a sample of volunteer patients, one month after the end of their follow-up, by a psychologist specializing in qualitative studies.
  The objective is to describe qualitatively the feasibility criteria for implementing the intervention according to the GUIDES checklist domains (A favorable context of use, appropriate content, a high-performance system, adequate implementation)
Other: Individual semi directive interview or r Focus Group with the primary care professional — Semi-structured individual interviews or focus groups with 24 primary care professionals will be conducted by a psychologist specializing in qualitative studies with a sample of volunteers, one month after the last patient's last visit to the center.
  The objective is to describe qualitatively the feasibility criteria for implementing the intervention according to the GUIDES checklist domains (A favorable context of use, appropriate content, a high-performance system, adequate implementation)

SUMMARY:
Primary care professionals (PCPs) are responsible for identifying patients who are eligible for all recommended screenings. Eligibility is difficult, given the number of screenings recommended by the French National Authority for Health (HAS), and the complexity of defining risk groups. When eligibility for one or more screenings is identified, the PCP informs the patient and can help him or her make the decision, considering his or her values and preferences.

Lack of information for patients and lack of time for PCPs are the main obstacles to prevention in primary care (PC). Another barrier identified is the lack of opportunity for patients who do not consult their PCP very often, as they are less likely to be approached for preventive interventions due to other more urgent reasons for consultation.

A Medical Decision Support System (MDSS) is a software application designed to be a direct aid to clinical decision-making, in which an inference engine matches individual patient characteristics with a computerized knowledge base or machine-learning algorithm to propose a risk assessment or adapted recommendations to the healthcare professional and/or patient.

The aim of the ADER-F research program is to support the development and evaluation of a complex intervention centred on the use of a MDSS called "Lianeli".

This complex intervention will ultimately contribute to structuring new consultations dedicated to prevention in general practice, by improving the physician's sense of self-efficacy in conducting the shared screening decision, and reducing the patient's decision-making conflict.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤74 years,
* Consultant to general practitioner,
* Without communication barriers in French, able to read and write
* Have signed the written consent form to participate in the study

Exclusion Criteria:

* Under legal protection (guardianship, curatorship, safeguard of justice or deprived of liberty)
* with a psychiatric pathology or disorder with impaired judgment, as determined by the GP
* Pregnant or breast-feeding
* Not affiliated to a social security scheme or not benefiting from a similar scheme
* Participating in another clinical study that may interfere with the ADER-F study-

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Lianeli SADM fully used | Within 60 days of the inclusion consultation
  The primary outcome is a composite criterion. This composite criterion is the proportion of patients with full use of the Lianeli SADM. A "yes" answer to the three following items defines full use of the Lianeli SADM:
  * Validation by the patient of their answers to the Lianeli health questionnaire (yes/no)
  * Validation by the general practitioner of the patient's responses to the Lianeli health questionnaire (yes/no)
  * Completion of the consultation dedicated to screening (yes/no)
Lianeli SADM fully used | Within 60 days of the inclusion consultation
  Proportion of patients included for whom the Lianeli SADM was fully used :
  Verification of the questionnaire by the GP (validate/not validated)
Lianeli SADM fully used | Within 60 days of the inclusion consultation
  Proportion of patients included for whom the Lianeli SADM was fully used :
  Dedicated screening consultation with the GP (done/not done)

SECONDARY OUTCOMES:
Feasibility criteria - GUIDES | Within 60 days of the inclusion consultation
  Describe quantitatively the feasibility criteria for the implementation of the ADER-F intervention according to the GUIDES checklist domains.
  The checklist GUIDES is the standard for evaluating indicators that promote the implementation of an CDS (computerized decision support) system based on clinical practice recommendations. According to this guide, indicators evenly distributed across four areas (a favorable context for use, an appropriate content, an effective system, a proper implementation) determine the success of an CDS system implementation. Questionnaire GUIDES consists of 12 items distributed across this four areas. Each item is scored using a 7-point Likert scale. Responses were code as follows : 1 for strongly disagree, 2 for disagree, 3 for somewhat disagree, 4 for undecided, 5 for somewhat agree, 6 for agree, 7 for strongly agree.
  The scores per domain are the average of the scores assigned to the various items comprising each domain (range 1 to 7). Domains with l
Feasibility crtiteria (Patient satisfaction questionnaire) | Within 30 days after the dedicated screening consultation with the GP
  Describe quantitatively the feasibility criteria for the implementation of the ADER-F intervention according to the GUIDES checklist domains using patient satisfaction questionnaire (12 items - 7-point Likert scale).
  The satisfaction questionnaire is interpreted according to the areas of the GUIDES Check List. According to this guide, 16 indicators, evenly distributed across 4 areas, determine the success of implementing a SADM (Simplified Access Management System). These four areas lead researchers to ensure that the context of use is favorable, the content appropriate, the system efficient, and the implementation adequate.
Feasibility criteria (Primary care professional satisfaction questionnaire) | Within 30 days after the dedicated screening consultation with the GP
  Describe quantitatively the feasibility criteria for the implementation of the ADER-F intervention according to the areas GUIDES checklist domains using primary care professional questionnaire (11 items - 7-point Likert scale)
Patient usability of Lianeli SADM | Within 30 days after the dedicated screening consultation with the GP
  Assessment of the Lianeli SADM user experience (patient and Primary care professional) using the SUS scale The System Usability Scale (SUS) is a questionnaire for measuring the usability of interactive systems, comprising ten items formulated in the form of affirmative sentences. For each sentence, users are asked to express their agreement or disagreement, using a 5-point Lickert scale.
  Assessment of the Lianeli SADM user experience (patient and Primary care professional) using the SUS scale The System Usability Scale (SUS) is a questionnaire for measuring the usability of interactive systems, comprising ten items formulated in the form of affirmative sentences. For each sentence, users are asked to express their agreement or disagreement, using a 5-point Lickert scale. The results of the SUS questionnaire are used to calculate the satisfaction score. This score ranges from 1 to 100. A score of 75 or above is generally considered "good," while a score between 50 and 75 is considered
Interprofessional use of the Lianeli SADM | Within 60 days of the inclusion consultation
  To assess the effect of interprofessional use of the Lianeli SADM on the primary endpoint.
  Interprofessional work will be defined as the collaboration of at least two healthcare professionals (including the general practitioner) with the patient as part of the ADER-F intervention
HLS-UE16 | Within 60 days of the inclusion consultation
  To assess the effect of patients' health literacy on the primary endpoint. Health literacy will be assessed using the HLS-EU16 (European Health Literacy Survey Questionnaire). This questionnaire comprises 16 questions using a 5-point Likert scale. The HLS-EU16 L scale assesses one dimension of health literacy in the general population. The French version of the HLS-EU-Q16 has acceptable psychometric properties.
  European Health Literacy Survey Questionnaire (Erreur dans proto - échelle Likert en 4 points) The results of the HLS-EU16 scale reveal the health literacy levels of the participants. Responses were coded as follows: 0 for "quite difficult" and "very difficult," and 1 for "quite easy" and "very easy." The total score, which ranges from 0 to 16, allows participants' health literacy to be classified into three levels: Inadequate (0-8), Problematic (9-12), Sufficient (13-16)
EPICES 11 | Within 60 days of the inclusion consultation
  EPICES : Assessment of Precarity and Health Inequalities in Health Examination Centers To assess the effect of patients' precariousness and health inequalities on the primary outcome.
  Health insecurity will be assessed using the EPICES scale. This questionnaire is an individual indicator of precariousness that considers the multidimensional nature of precariousness. It consists of 11 binary yes/no questions. The answer to each question is assigned a coefficient, and the sum of the 11 answers gives the EPICES score. The score is continuous, ranging from 0 (absence of precariousness) to 100 (maximum precariousness). A single score of 30.17 is considered relevant.
Organized cancer screenings (breast, cervical and colorectal) | Within 60 days of the inclusion consultation
  The proportion of patients for whom the intervention is likely to improve participation in the three organized cancer screenings (colorectal, breast, cervical) will be assessed within the population of patients identified as eligible for at least one of the three organized screenings (previous examination performed within a timeframe greater than the recommended timeframe, or never performed) by the proportion of patients who attended the dedicated screening consultation within 60 days of the inclusion consultation.
Individual cancer screening | Within 60 days
  The proportion of patients for whom the intervention is likely to improve participation in opportunistic cancer screening will be assessed within the population of patients identified as eligible for at least one of the opportunistic cancer screenings (high-risk colorectal cancer, high-risk breast cancer, high-risk stomach cancer - previous examination performed within a timeframe greater than the recommended timeframe or never performed) by the proportion of patients who attended the dedicated screening consultation within 60 days of the inclusion consultation.
Feasibility criteria - metadata | Within 60 days of the inclusion consultation
  Describe quantitatively the feasibility criteria for the implementation of the ADER-F intervention from Lianeli usage metadata

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Cabinet médical, Belley
  - Cabinet médical, Beynost
  - CSCP - Centre de Santé Communautaire et Planétaire, Bron
  - Cabinet médical, Craponne
  - MSP, Crêches-sur-Saône
  - Maison de santé Gleizé Epinay, Gleizé
  - Groupe Médical Claude Bernard, LArbresle
  - Cabinet médical, Lyon
  - Maison de Santé Beauvisage, Lyon
  - Cabinet médcial, Saint-Pierre-la-Palud
  - MSP du Tissage, Tignieu
  - Cabinet médical, Villeurbanne
  - Maison de Santé Clos Caroline, Villeurbanne